CLINICAL TRIAL: NCT06917729
Title: Responses on Arterial Stiffness and Cardiac Vagal Modulation to Breathing Exercises Through the Use of CardioBreath Application in Hypertension and Pre Hypertension; a Randomized Clinical Trial
Brief Title: Breathing Exercises of CardioBreath Application on Autonomic and Vascular Function in Hypertension
Acronym: CardioBreath
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Janaina Pinheiro, Nurse, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6131/24; 7.323.318 (Other: Organizational Ethical Comitee)
Record Dates: First submitted 2025-03-18; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Pre Hypertension
Keywords: Hypertension; Breathing Exercises; Blood Pressure
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (1:1) to intervention via the website www.randomization.com :Group 1-Group with intervention and Group 2-Non- intervention group (control). After randomization, participants will be instructed on how their group's intervention will work, and will also receive the instruments and equipment to carry out the intervention, at no personal cost.
  The sessions used will be the Prescription, based on data from the users' profile, including the Spontaneous Respiratory Rate (SRR) as the basis for prescribing the exercises, the relaxation section, and the Victorious section, where the user achieves mastery over his/her breathing. The same will be installed free of charge on the participant's cell phone . In group 2 (without intervention), participants will receive teaching material based on the lessons from the CardioBreath and after the time of intervention they will receive freely the Cardiobreath application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CardioBreath Application (Active Comparator): Lessons in the CardioBreath app are based on the breathing techniqueUjjayi Pranayama(Victorious breathing), which uses the narrowing of the glottis through a soft noise in the throat to prolong the two phases of breathing. The sessions used for the intervention will be the Prescription, based on data from the users' profile, including the Spontaneous Respiratory Rate (SRR) as the basis for prescribing the exercises, the relaxation section, which aims to deeply relax the respiratory muscles and others, and the Victorious section, where the user achieves mastery over his/her breathing.
  Interventions: Other: CardioBreath
- Control (Sham Comparator): Participants will receive graphic material based on the contents of cardioBreath Application, with instructions to be aware of their breath , control it towards lower rates by increasing respiratory phases through ujjayi pranayama
  Interventions: Other: CardioBreath

INTERVENTIONS:
Other: CardioBreath — Twice a day for ten minutes,5 days during the week CardioBreath app will be based on Prescription section , using breathing technique Ujjayi Pranayama, based on spontaneous respiratory rate of users, gamified to induce the user to improve performance of the exercises reducing the exercises respiratory exercises
  Other Names: CardioBreath Application

SUMMARY:
Hypertension is one of the greatest public health challenges, affecting more than one billion people worldwide and representing a significant financial and public health burden. It is responsible for a high number of cardiovascular events, such as heart attacks and strokes. Although pharmacological treatment is effective, non-pharmacological interventions are essential for the sustainable management of blood pressure, especially in its early stages. Respiratory exercises have shown potential in reducing blood pressure and improving cardiac vagal modulation, promoting cardiovascular health benefits.

This study aims to evaluate the effectiveness of guided respiratory exercises using the CardioBreath app in improving vagal modulation and reducing arterial stiffness in adults with prehypertension or hypertension over six weeks. This is a randomized clinical trial involving adults with prehypertension or hypertension, divided into intervention and control groups. The intervention group will use CardioBreath to perform daily breathing exercises, with weekly remote monitoring. Assessments will include heart rate variability parameters, baroreflex sensitivity, pulse wave velocity, and quality of life.

It is expected that the use of the app will significantly improve vagal modulation and arterial stiffness, demonstrating the potential of this intervention for the non-pharmacological management of hypertension. The use of CardioBreath may offer an accessible and effective alternative for blood pressure control, with the potential to be integrated into public health programs focused on low-cost, highly accessible interventions for the prevention and management of hypertension.

DETAILED DESCRIPTION:
Systemic Arterial Hypertension (SAH) affects 1.33 billion people globally, representing 10% of global health costs. In the US, a study published in 2019 estimated that annual spending due to hypertension was $56 billion. According to the Surveillance Survey of Risk and Protective Factors for Chronic Diseases by Telephone Survey (Vigitel), carried out in 2021 and with a report published in 2022, the frequency of adults (18 years or older) in Brazilian capitals who reported a medical diagnosis of hypertension was 26.3%. This represents an increase in relation to the data from 2011, when the percentage was 24.3%. Hypertension is the main risk factor for events such as Acute Myocardial Infarction (AMI) and Stroke (CVA). The mortality rate due to hypertension in Brazil reached the highest value in the last ten years, with 18.7 deaths per 100,000 inhabitants in 2021 .

The 2024 European Society of Cardiology (ESC) Guideline on the management of elevated blood pressure (BP) and hypertension presents significant changes from previous versions. The new title reflects the understanding of cardiovascular risk as a continuous spectrum, emphasizing the importance of accurate BP measurement, recommending the use of validated devices, standardized techniques, and out-of-office measurement.

Treatment strategies include lifestyle interventions and drug therapy, with an emphasis on lower BP targets and combination therapy from the outset, addressing the management of hypertension in specific populations, such as women, the elderly, patients with Chronic Kidney Disease (CKD) and Diabetes Mellitus (DM). Resistant and secondary hypertension are also discussed, with recommendations for diagnosis and treatment. Psychosocial aspects, such as communication of diagnosis and adherence to treatment, are highlighted. Self-care and BP monitoring are encouraged, with the caveat that evidence for digital tools is still limited, recommending the importance of a patient- centered approach and shared decision-making. Lifestyle change is considered an essential component in the management of high blood pressure and hypertension.

Within this context, the need to control blood pressure values is expressed in order to reduce risks and contain the progression of the pathology, the inclusion of non-pharmacological approaches becomes imperative. Referring to the genesis of hypertension, there is an imbalance in the Autonomic Nervous System (ANS), which presents a sustained increase in sympathetic neural activity and a reduction in vagal modulation, implying a reduction in

baroreflex sensitivity, the heart's beat-to-beat blood pressure regulatory mechanism, generating a sustained increase in blood pressure (BP) values and the establishment of hypertension.

The vast literature and studies by this research group indicate that slow and deep breathing exercises reduce blood pressure levels, increasing cardiac vagal modulation, with the potential to restore baroreflex sensitivity. This low-cost non- pharmacological intervention can be used for both prevention and treatment of hypertension and does not pose additional risks.

A study by this research group also demonstrated that postmenopausal hypertensive women who practiced a yoga and stretching protocol in association with a breathing technique for 12 weeks obtained a reduction in resting heart rate (HR) and arterial stiffness assessed by Pulse Wave Velocity (PWV). Stiffness of the central arteries is considered an early predictor of risk when PWV> 10 m/s. For each increase of 1 m/s in PWV, there is an increase in the risk of cardiovascular death, cardiovascular event and death from all causes of around 14-15% .

Breathing exercises are an effective non-pharmacological intervention for the treatment and prevention of pre-hypertension and hypertension. A study evaluated the impact of breathing exercises in hypertensive individuals and demonstrated improvement in chest expansion, reduction in blood pressure and increase in heart rate variability, a reliable index of vagal modulation . Breathing exercises, called pranayamas, can influence physiological states and psychological.

The study, led by Dr. Maria Claudia Irigoyen, compared yoga practitioners with healthy sedentary individuals and found that yoga practitioners had higher maximal expiratory pressure (MEP), greater abdominal and thoracic expansion, and significantly lower resting heart rates. These results suggest that breathing exercises may have a positive impact on blood pressure and cardiovascular health .

Furthermore, the applicability of slow breathing exercises also favors the improvement of mental and cognitive health, which can facilitate lifestyle changes, especially the adoption of a more appropriate diet and the inclusion of regular exercise, in addition to promoting self-knowledge and self-monitoring.

In the context of health, the use of information and communication technologies has stood out as a means of democratizing and expanding access to knowledge, being an important resource for health care, helping both professionals and patients/users (Casaeset al., 2021). Recently, a review on the growing trend of using mobile applications related to healthy lifestyles pointed to more than 5,400 applications available for use, indicating the digital medium as a potential tool for promoting healthy habits and preventing chronic diseases, in addition to enhancing public health initiatives.

Considering the clinical underutilization of breathing interventions, and in order to increase their accessibility, the CardioBreath® App was created, developed and implemented. Structured through the union of theoretical principles of research carried out with slower respiratory rates (RR) on blood pressure and cardiac vagal modulation at the Institute of Cardiology of RS/Universitary Foundation of Cardiology (ICFUC-RS) and the practical principles of Yoga, the app was designed by Prof. Dr. Cláudia Fetter and collaborators and is available on Google Play and AppStore (www.cardiobreath.com).

The application prescribes, guides, monitors and rewards the practice of breathing exercises through a guided audiovisual system, benefiting the user through its simplicity, availability and efficiency. Through the acquisition of biological signals, heart rate (HR) and spontaneous respiratory rate (SRR), the user receives their exercise prescription and can monitor their results. Along with the "Prescription" section, the "Relaxation" section represents the user's initial contact, who is gamified and encouraged to progress towards mastery over breathing in the "Victors" section. Given the above, the objective of the present study is to evaluate, diagnose and recommend actions to individuals with pre-hypertension and hypertension through a Randomized Clinical Trial using the CardioBreath application for 6 weeks on autonomic and vascular outcomes.

JUSTIFICATION

Systemic Arterial Hypertension (SAH) affects one in three adults around the world, and the number of people living with hypertension (blood pressure greater than or equal to 140/90 mmHg) doubled between 1990 and 2019, rising from 650 million to 1.3 billion (UN, 2022).

The alarming prevalence of hypertension reaches around 27.9% of the Brazilian population, with a higher medical diagnosis among women (29.3%) compared to men.

reach 26.4% in the 27 Brazilian capitals. The data indicate that the frequency increases with age in the population and low rates of control of BP values (Brazil, 2023).

The publication in 2023 of the first report by the World Health Organization (WHO) corroborates the critical global effects of hypertension, including recommendations for its control. Approximately four out of five individuals diagnosed with hypertension do not receive treatment that is appropriate for their case. Every hour we have data from more than 1,000 individuals who die as a result of related complications. It is understood that countries with the possibility of expanding coverage and guiding treatment with associated non-pharmacological measures will be responsible for preventing 76 million deaths between 2023 and 2050.

In accordance with the recommendations of cardiology guidelines related to lifestyle changes, especially the adoption of a healthier diet with reduced sodium, regular exercise and stress management, they demonstrate the need to implement non-pharmacological strategies in the monitoring of these patients.

Considering the underutilization of slow breathing exercises applied in the control of chronic diseases such as hypertension, this study proposes the use of the CardioBreath application, developed together with the Clinical Research Laboratory (LIC) of the Institute of Cardiology: University Foundation (ICFUC), as a strategy for changingmindsetfor individuals with pre-hypertension and hypertension.

The availability of the application and the gradual inclusion of the practice of slow breathing exercises may represent an advance in the approach with these patients to reverse chronic sedentary lifestyle conditions, in addition to the possibility of improving psycho- emotional aspects such as anxiety and dietary control.

This study connects with the United Nations Sustainable Development Goals established for 2030, more specifically in objective 3 - Good Health and Well-being and in objective 9 - Industry, innovation and infrastructure, specifically including sub-item 9.b, which supports technological development, research and national innovation in developing countries, ensuring a conducive policy environment for, among other things, industrial diversification and value addition to commodities and in objective 9.5, providing for the strengthening of scientific research, improving the technological capabilities of industrial sectors in all countries, particularly developing countries, encouraging innovation and substantially increasing the number of workers and public and private spending on research and development.

ELIGIBILITY:
Inclusion Criteria:

* BP>130mmHg X 80mmHg or previous medical diagnosis of pre- hypertension or hypertension

Exclusion Criteria:

* use of beta-blockers
* drugs that depress the central nervous system
* clinical conditions that prevent participation after evaluation by the team
* individuals without a cell phone or tablet (which would make the proposed study unfeasible

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Cardiac Vagal Modulation | At baseline and after six weeks
  Cardiac vagal modulation obtained by the heart rate variability (HRV) in frequency domain conducted in the Finometer System, with a finger installed in the middle finger of the right hand of the patient, with a continuous peripheric blood pressure signal, collected with the subjects in rest position, in a room with light and temperature controlled. Baseline data is collected for ten minutes immediatly after the Finometer calibration.Following this, the subject will undergo slow breath exercise throught the CardoBreath application for five minutes, and afterward a new sequency of ten minutes of data collection. The signals are ransformed from a analogic-to-digital sequency, and analysed by Cardiseries software. Vagal modulation will be considered the high frequency (HF) band of the frequency domain analysis, between 0,15 to 0,4 Hz.

SECONDARY OUTCOMES:
Pulse wave velocity | At baseline and after six weeks
  Pulse wave velocity (PWV) is obtained by the oscilometric method, dividing the carotid- femoral distance by the travel time of the systolic wave. PWV will be measured by Arteris equipment in a seated position, at rest, in an environment with controlled temperature and lighting, with the cuff fitted to the left upper limb. Before the collection, the individual must empty their bladder and during the data collection, they must remain at rest for the measurement, in a quiet environment, with controlled temperature (± 23 ° C) and lighting. The device will perform 4 blood pressure measurements, the first measurement will be discarded and the other three will be analyzed by the MAPA's software to calculate the PWV.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia do RioGrande do Sul, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No